CLINICAL TRIAL: NCT06835998
Title: The Effect of Stress Ball Use on Stress, Sleep Quality, and Comfort Levels in Hemodialysis Patients: A Randomized Controlled Study
Brief Title: The Effect of Stress Ball Use on Stress, Sleep Quality and Comfort Levels
Acronym: Stress Ball
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Ayse Vicdan, Associate professor, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MuglaSitkiKocmanUniversity
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Hemodialysis
Keywords: Stress Ball; Sleep Quality; Comfort Levels; Hemodialysis Patients
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: randomized controlled, parellel
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patients involved in the study, the researcher collecting the pre-test and post-test data, and the statistician evaluating the data were not informed about the group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stress ball (Experimental): the stress ball intervention was initiated. Before starting, the researcher provided instructions and demonstrations on how to use the stress ball, allowing then the patients to practice. The stress ball intervention was administered during the second hour of the hemodialysis session when patients were most comfortable. Patients were instructed to squeeze the stress ball once, counting internally as "1-2-3" with each squeeze. The stress ball intervention was administered three times weekly during hemodialysis sessions for 15 minutes each session, totaling 12 sessions for a period of four weeks. Throughout the intervention, patients were observed by the same researcher.
  Interventions: Other: stress ball
- Control (No Intervention): No intervention will be made to the contro group, only data will be collected at the same time as the study group.

INTERVENTIONS:
Other: stress ball — the stress ball intervention was initiated. Before starting, the researcher provided instructions and demonstrations on how to use the stress ball, allowing then the patients to practice. The stress ball intervention was administered during the second hour of the hemodialysis session when patients were most comfortable. Patients were instructed to squeeze the stress ball once, counting internally as "1-2-3" with each squeeze. The stress ball intervention was administered three times weekly during hemodialysis sessions for 15 minutes each session, totaling 12 sessions for a period of four weeks. Throughout the intervention, patients were observed by the same researcher.
  Arms: stress ball

SUMMARY:
This study was conducted to determine the impact of stress ball use on stress, sleep quality, and comfort levels in hemodialysis patients.

DETAILED DESCRIPTION:
The study population consisted of patients undergoing hemodialysis treatment in the hemodialysis unit of a training and research hospital located in western Türkiye between February 19, 2024, and April 19, 2024 (N=90). The study sample included a total of 60 patients (30 in the experimental group and 30 in the control group), selected through randomization from those who met the research criteria and agreed to participate. During the study, two patients from the experimental group and one patient from the control group were excluded from the study due to health issues that prevented them from using the stress ball. The study was conducted with a total of 57 patients (28 in the experimental group and 29 in the control group).

ELIGIBILITY:
Inclusion Criteria:

* participants had to be volunteers
* aged 18 years and older,
* undergoing hemodialysis treatment for at least six months,
* attending hemodialysis sessions three times a week,
* not having any conditions that would impede the use of a stress ball.

Exclusion Criteria:

* individuals who refused to participate in the study,
* those undergoing hemodialysis for less than six months,
* patients attending hemodialysis sessions twice a week,
* individuals with health problems that prevented them from using a stress ball.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Stress evaluated using the Perceived Stress Scale | Change from before implementation and 4th week of practice
  The obtainable total score from the scale ranges from 0 to 56, with higher scores indicating a greater perception of stress
Sleep quality ewaluated the Pittsburgh Sleep Quality Index | Change from before implementation and 4th week of practice
  The sum of the scores from these seven components yields the total PSQI score, which ranges from 0 to 21. Individuals with a total score of 5 or lower are classified as having 'good" sleep quality, while those with a score above 5 are classified as having "poor" sleep quality.
Comfort evaluated using Hemodialysis Comfort Scale Version II | Change from before implementation and 4th week of practice
  The total score obtained from the scale ranges from 26 to 130, with higher scores indicating greater comfort levels.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Kacaroglu Vicdan, Associate Professor, Principal Investigator — Muğla Sıtkı Koçman Universty; Dilek Dilek Gibyeli Genek, Assisstant Professor, Study Chair — Muğla Sıtkı Koçman Universty
Locations (1):
- Turkey, Muğla Sıtkı Koçman University, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All information about the study can be shared
Supporting Information: Study Protocol, ICF
Time Frame: 14 february 2025 -14 february 2026
Access Criteria: All information about the study can be shared